CLINICAL TRIAL: NCT04479176
Title: Comparison of Temperature and Pain Changes Between the Drip and Topical Methods of Administering the Transnasal Sphenopalatine Ganglion Block
Brief Title: Comparison of Two Methods of Transnasal Sphenopalatine Ganglion Block
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Bum Choi, Assistant Professor, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-MDB-20-565
Record Dates: First submitted 2020-07-15; First posted 2020-07-21 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Sphenopalatine Ganglion Block

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Drip-method group: Transnasal SPGB was performed by a single pain clinician. After the patient was placed in a supine and neck-extended position, 2 mL of 2% mepivacaine was placed in a syringe connected to a 16-gauge Angiocath sheath. The sheath of the Angiocath was inserted through the nostril, and 2% mepivacaine was dripped into the nostrils with the patient in a supine position. The mepivacaine drip on the nasal pharynx was maintained for 10 min. A drip of 2% mepivacaine was delivered to the nostril, where the pain was dominant. In cases of bilateral pain, mepivacaine drip was administered to both nostrils.
  Interventions: Procedure: Transnasal Sphenopalatine Ganglion Block
- Topical-method group: Transnasal SPGB was performed by a single pain clinician. The posture was the same as that in the drip method. A cotton tip applicator soaked with 2% mepivacaine was inserted vertically into the nostril. After the cotton tip applicator made contact with the posterior wall of the middle turbinate, the cotton tip applicator was fixed for 10 min. A cotton tip applicator was inserted into the nostril, where the pain was dominant. In cases of bilateral pain, two applicators were inserted into both nostrils.
  Interventions: Procedure: Transnasal Sphenopalatine Ganglion Block

INTERVENTIONS:
Procedure: Transnasal Sphenopalatine Ganglion Block — In transnasal approach, several authors described the traditional technique using sterile 10cm cotton tipped applicators that are dipped in the chosen anesthetic and then advanced along the superior border of the middle turbinate, until it reaches the posterior wall of the nasopharynx. Some other techniques had described dripping one or two ml of the anesthetics into the nostril.

SUMMARY:
The transnasal sphenopalatine ganglion block(SPGB) is administered to patients with facial or head and neck pain. In the transnasal approach, the drip and topical methods are frequently used. We compared facial temperatures and VAS after transnasal SPGB.

DETAILED DESCRIPTION:
The objective of this study was to compare facial temperatures and visual analogue scale (VAS) between drip method and topical method of transnasal sphenopalatine ganglion block (SPGB).

The transnasal SPGB is administered to patients with facial or head and neck pain. In the transnasal approach, the drip and topical methods are frequently used. We compared facial temperatures and VAS after transnasal SPGB.

Medical records of 74 patients who visited the pain clinic and underwent transnasal SPGB were retrospectively reviewed. A total of 156 transnasal SPGB were performed. The patients were divided into the drip-method and topical-method groups. Facial temperatures were measured in six areas of the right and left forehead, maxilla, and mandible before and 30 min after completion of the transnasal SPGB. Temperatures were compared before and 30 min after SPGB in each group and between the two groups. VAS scores were compared at same times of SPGB in each group and between the two groups.

ELIGIBILITY:
Inclusion Criteria:

(1) age over 20 years ; (2) head and neck pain; (3) pain score > 4 on the VAS in the head and neck; and (4) having undergone a transnasal SPGB and having had facial temperatures measured.

Exclusion Criteria:

(1) patients with a history of head and neck surgery, (2) treatment with a vasodilator or vasoconstrictor, (3) contraindication to treatment using a transnasal approach, (4) clinically significant systemic disease or any reduced organ failure, and (5) missing data.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who visited pain clinic of Ajou university hospital, and a total of 74 patients who be performed transnasal sphenopalatine ganglion block
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Facial temperatures | Before, and 30 minutes after completion of transnasal sphenopalatine ganglion block
  Facial temeratures changes after transnasal SPGB
Visual analogue scale(VAS) | Before, and 30 minutes after completion of transnasal sphenopalatine ganglion block
  11 points pain scale score from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Kim, Study Chair — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, Gyunggi, South Korea

IPD SHARING:
Plan to Share IPD: No